CLINICAL TRIAL: NCT00594984
Title: A Blinded, Randomized, Phase 1/2 Study of Brivanib Alaninate vs Placebo in Combination With Erbitux and Irinotecan K-Ras Wildtype Subjects With Metastatic Colorectal Cancer
Brief Title: Phase I/II Combination With Irinotecan- Erbitux
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA182-025; 2007-005097-31
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Colorectal Cancer (MCRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan; brivanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 - Phase 1 (Active Comparator): Cetuximab + Irinotecan + Brivanib
  OR
  Cetuximab + Irinotecan + Brivanib Placebo
  Interventions: Drug: Cetuximab; Drug: Irinotecan; Drug: Brivanib; Drug: Brivanib Placebo
- Arm 2 - Phase 2 (Placebo Comparator): Cetuximab + Irinotecan + Brivanib
  OR
  Cetuximab + Irinotecan + Brivanib Placebo
  Interventions: Drug: Cetuximab; Drug: Irinotecan; Drug: Brivanib; Drug: Brivanib Placebo

INTERVENTIONS:
Drug: Cetuximab — IV solution, IV, QW, 400 mg/m2 X 1, followed by 250mg/m2, until progression
  Other Names: Erbitux; BMS-564717
Drug: Irinotecan — IV solution, IV, Q3W, 350 mg/m2, until progression
Drug: Brivanib — Oral, Tablet, QD, (200 mg, 400 mg, 600 mg, 800 mg dose escalation) until progression
  Arms: Arm 1 - Phase 1
Drug: Brivanib — Oral, Tablet, QD, MTD determined in Arm 1, Phase 1, until progression
  Arms: Arm 2 - Phase 2
Drug: Brivanib Placebo — Oral, tablet, QD, until progression

SUMMARY:
Part 1: To define the recommended dose of brivanib that can be safely administered in combination with Erbitux (Cetuximab) and irinotecan to subjects with advanced metastatic colorectal cancer (MCRC)

Part 2: To compare median duration of progression free survival (PFS)

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven MCRC
* Prior irinotecan allowed
* Prior Erbitux allowed

Exclusion Criteria:

* No prior brivanib
* No prior combination of irinotecan with Erbitux
* No secondary malignancies
* No anti-coagulation therapy
* No prior history of blood clots requiring anti-coagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics and markers of exploratory coagulation pathways will be conducted during this trial | PK C1D1-C2-D3, biomarker throughout the study
Safety and tolerability of interventions will be collected | throughout the study on Part II

SECONDARY OUTCOMES:
Efficacy on tumor progression and progression free survival will be collected on all enrolled subjects | throughout the study on Part II

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- United States (4):
  - Usc/Norris Comprehensive Cancer Center Hospital, Los Angeles, California
  - Usc/Norris Comprehensive Cancer Center, Los Angeles, California
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Washington University, St Louis, Missouri
- Local Institution, Buenos Aires, Buenos Aires, Argentina
- Local Institution, Odense C, Denmark
- Italy (2):
  - Local Institution, Meldola Fc
  - Local Institution, Milan
- Local Institution, Seoul, South Korea
- Local Institution, Madrid, Spain
- Sweden (2):
  - Local Institution, Stockholm
  - Local Institution, Uppsala

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx